CLINICAL TRIAL: NCT00472121
Title: The Precision and Arm-to-Arm Variation og Mechanomyography and Acceleromyography for Monitoring the Neuromuscular Block During Anesthesia, A Randomized Controlled Study
Brief Title: The Precision and Arm-to-Arm Variation of Mechanomyography and Acceleromyography for Monitoring of Neuromuscular Block
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Other Study IDs: MMG-MMG
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Last update posted 2008-04-18 (Estimated); Status verified 2008-04

CONDITIONS: Neuromuscular Blockade

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: AMG
  Interventions: Device: TOF-Watch SX (neuromuscular monitor)
- 2: MMG
  Interventions: Device: TOF-Watch SX (neuromuscular monitor)

INTERVENTIONS:
Device: TOF-Watch SX (neuromuscular monitor) — The variation between arms (dominant or non-dominant) when monitored with the same method on both arms

SUMMARY:
The purpose of the study is the examine the precision of acceleromyography and mechanomyography during recovery from a neuromuscular blocking agent and to examine whether there is any difference in monitoring block at the dominant or non-dominant arm. Our hypothesis is that there is no significant difference in neither the precision nor the level of block in the contralateral arms.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* General anesthesia >1 hour
* Surgery in supine position w. possibility of monitoring the neuromuscular block at both arms (n. ulnaris stimulation/thumb response)
* Written informed content

Exclusion Criteria:

* Neuromuscular disorders, hepatic and renal dysfunction
* Medication expected to interfere with the neuromuscular blocking agent
* Allergy to any medication used during anaesthesia
* Body weight less or exceeding 20% of ideal body weight
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2007-05; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Precision at the contralateral arms using the average residual coefficient of variation over subsequent linear regressions (detrending) over time

SECONDARY OUTCOMES:
Bias and limits of agreement between control TOF, reappearance of T1, T2, T3, T4
T1 height at reappearance of T1-T4
Time to T1=25%
Interval 25-75%
Time to TOF 0.9 and 1.0 with and without normalization
Time to stable T1 and stable TOF

CONTACTS AND LOCATIONS:
Overall Officials: Casper C Kjær, MD, Principal Investigator — Dep. of anaesthesia 4231, Rigshospitalet
Locations (1):
- Dep. of Anaesthesia, Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Claudius C, Skovgaard LT, Viby-Mogensen J. Arm-to-arm variation when evaluating neuromuscular block: an analysis of the precision and the bias and agreement between arms when using mechanomyography or acceleromyography. Br J Anaesth. 2010 Sep;105(3):310-7. doi: 10.1093/bja/aeq162. Epub 2010 Jun 30. PMID 20595196